CLINICAL TRIAL: NCT06219967
Title: Does a Soft Drink Mixture Improve Tolerance of Activated Charcoal in the Adult Poisoned Patient Without Affecting Efficacy: A Randomized Crossover Trial
Brief Title: Does a Soft Drink Mixture Improve Tolerance of Activated Charcoal in the Adult Poisoned Patient Without Affecting Efficacy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Principal Investigator, Michael Keenan, Assistant Professor Emergency Medicine, State University of New York - Upstate Medical University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1783698-11
Record Dates: First submitted 2024-01-02; First posted 2024-01-23 (Actual); Results first posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Overdose
MeSH Terms: conditions — Drug Overdose | interventions — Charcoal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Activated charcoal with cola (Experimental)
  Interventions: Drug: Activated Charcoal
- Activated charcoal (Active Comparator)
  Interventions: Drug: Activated Charcoal

INTERVENTIONS:
Drug: Activated Charcoal — Activated charcoal alone
  Arms: Activated charcoal
Drug: Activated Charcoal — Activated charcoal mixed with cola
  Arms: Activated charcoal with cola

SUMMARY:
Activated charcoal (AC) is an established, effective means of gastrointestinal decontamination. Providers give it to patients who have ingested something that is thought to be potentially poisonous to prevent it from being absorbed. However, one limitation to its use is palatability of the AC for the patient, potentially limiting how much, if any, is taken.

Other studies have suggested that mixing AC with various substances improves the rating on various scales (taste, etc). An important question is whether mixing the AC with other substance effects the ability of the AC to bind to xenobiotic in the gut. This small study investigates whether mixed cola with charcoal affected its ability to prevent the absorption of acetaminophen. It also performs a survery to see if participants preferred the AC-cola mixture. The investigators hypothesize that the AC will be equally as effective with cola as without. The investigators also hypothesize that participants will prefer the AC-cola mixture.

ELIGIBILITY:
Inclusion Criteria:

* No self-reported history of any hepatic, gastrointestinal, or renal disease
* No self-reported history of alcohol or substance use disorder
* No daily prescribed medications
* Weight between 60-93 kg

Exclusion Criteria:

* pregnant,
* imprisoned
* allergy or intolerance to acetaminophen or gluten

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2023-01-04 (Actual); Primary Completion 2023-03-14 (Actual); Study Completion 2023-03-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- SUNY Upstate Medical University Clinical Research Unit, Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 5 participants were screened for eligibility between January 4, 2023 and February 27, 2023.
Pre-assignment Details: All 5 screened participants met criteria for involvement in the study. Participants were randomized to receive either the charcoal or charcoal-cola mixture first, then, after at least 7 days between each session, the participants returned to complete the other arm of the study.
Groups:
- Activated Charcoal With Cola First, Then Activated Charcoal Alone: Participants in this arm conducted the protocol with 50 g activated charcoal mixed with 240 mL of cola on study day 1. After a minimum of a 7 day washout period, they returned and repeated the protocol with 50 g activated charcoal alone.
- Activated Charcoal Alone First, Then Activated Charcoal With Cola: Participants in this arm conducted the protocol with 50 g activated charcoal alone on study day 1. After a minimum of a 7 day washout period, they returned and repeated the protocol with 50 g activated charcoal mixed with 240 mL of cola.
Period: Study Day 1
Arm/Group | Activated Charcoal With Cola First, Then Activated Charcoal Alone | Activated Charcoal Alone First, Then Activated Charcoal With Cola
Started | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0
Period: Washout (at Least 7 Days)
Arm/Group | Activated Charcoal With Cola First, Then Activated Charcoal Alone | Activated Charcoal Alone First, Then Activated Charcoal With Cola
Started | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0
Period: Study Day 2
Arm/Group | Activated Charcoal With Cola First, Then Activated Charcoal Alone | Activated Charcoal Alone First, Then Activated Charcoal With Cola
Started | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Activated Charcoal With Cola First: Participants received activated charcoal mixed with cola, then received activated charcoal alone
- Activated Charcoal Alone First: Participants received activated charcoal alone, then received activated charcoal mixed with cola
- Total: Total of all reporting groups
Arm/Group | Activated Charcoal With Cola First | Activated Charcoal Alone First | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Continuous [Mean (Full Range); unit: years] | 34 [31 to 36] | 29 [28 to 30] | 32 [28 to 36]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Absorption of Acetaminophen as Indicated by Area Under the Curve
Description: Measure of the area under the curve of the acetaminophen concentration vs time curve. Values obtained at 0, 15, 30, 45, 60, 75, 90, 120, 180, and 240 minutes were used to produce the curve
Time Frame: 240 minutes
Measure: Mean (95% Confidence Interval); unit: mcg*min/mL
Groups:
- Activated Charcoal With Cola: Activated charcoal mixed with cola
- Activated Charcoal Without Cola: Activated charcoal without cola (charcoal by itself)
Arm/Group | Activated Charcoal With Cola | Activated Charcoal Without Cola
Number analyzed (Participants) | 5 | 5
mcg*min/mL | 3566 [1390 to 5742] | 3335 [2573 to 4098]

2. Primary Outcome: Maximum Concentration Acetaminophen
Description: Maximum concentration of acetaminophen (mcg/mL)
Time Frame: 240 minutes
Measure: Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | Activated Charcoal With Cola | Activated Charcoal Without Cola
Number analyzed (Participants) | 5 | 5
mcg/mL | 33 [7 to 59] | 29 [20 to 37]

3. Primary Outcome: Time to Maximum Concentration of Acetaminophen
Description: Time of maximum concentration of acetaminophen (minutes)
Time Frame: 240 minutes
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Activated Charcoal With Cola | Activated Charcoal Without Cola
Number analyzed (Participants) | 5 | 5
minutes | 51 [30 to 72] | 66 [56 to 76]

4. Secondary Outcome: Appeal of Charcoal Mixture
Description: Participant rating of the appearance of charcoal mixture on a scale of 0 to 10, with 10 being the most appealing and 0 being the least appealing
Time Frame: 5 minutes
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Activated Charcoal With Cola | Activated Charcoal Without Cola
Number analyzed (Participants) | 5 | 5
score on a scale | 4.6 [3.5 to 5.7] | 2.8 [1.0 to 4.6]

5. Secondary Outcome: Smell of Charcoal Mixture
Description: Participant rating of the smell of charcoal mixture on a scale of 0 to 10, with 10 being the most appealing and 0 being the least appealing
Time Frame: 5 minutes
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Activated Charcoal With Cola | Activated Charcoal Without Cola
Number analyzed (Participants) | 5 | 5
units on a scale | 5.8 [2.7 to 8.9] | 6.4 [3.0 to 9.8]

6. Secondary Outcome: Flavor of Charcoal Mixture
Description: Participant rating of the flavor of charcoal mixture on a scale of 0 to 10, with 10 being the most appealing and 0 being the least appealing
Time Frame: 5 minutes
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Activated Charcoal With Cola | Activated Charcoal Without Cola
Number analyzed (Participants) | 5 | 5
score on a scale | 5.8 [4.2 to 7.4] | 3.0 [0.0 to 6.3]

7. Secondary Outcome: Texture of Charcoal Mixture
Description: Participant rating of the texture of charcoal mixture on a scale of 0 to 10, with 10 being the most appealing and 0 being the least appealing
Time Frame: 5 minutes
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Activated Charcoal With Cola | Activated Charcoal Without Cola
Number analyzed (Participants) | 5 | 5
score on a scale | 4.4 [2.3 to 6.5] | 2.8 [1.2 to 4.4]

8. Secondary Outcome: Overall Appeal of Charcoal Mixture
Description: Participant rating of the overall appeal of charcoal mixture on a scale of 0 to 10, with 10 being the most appealing and 0 being the least appealing
Time Frame: 5 minutes
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Activated Charcoal With Cola | Activated Charcoal Without Cola
Number analyzed (Participants) | 5 | 5
score on a scale | 4.4 [3.7 to 5.1] | 3.2 [0.0 to 6.4]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded on study days 1 and 2, for the duration of the study day (Entirety of each study day approximately 240 minutes)
Groups:
- Activated Charcoal With Cola: Participants received activated charcoal mixed with cola (either first or after a
- Activated Charcoal Alone: Activated charcoal alone first
Arm/Group | Activated Charcoal With Cola | Activated Charcoal Alone
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-28): https://cdn.clinicaltrials.gov/large-docs/67/NCT06219967/Prot_SAP_002.pdf
  • Informed Consent Form (2022-11-28): https://cdn.clinicaltrials.gov/large-docs/67/NCT06219967/ICF_001.pdf